CLINICAL TRIAL: NCT00287833
Title: Phase I Single Dose Safety and Pharmacokinetic Study of Bowman Birk Inhibitor Concentrate, Delivered as an Orange Juice Suspension to Healthy Male Volunteers Between 18 and 65 Years of Age
Brief Title: Bowman-Birk Inhibitor Concentrate in Preventing Cancer in Healthy Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: NCI-2011-01479; UPCC-706366; N01-CN-25118; CDR0000429594
Record Dates: First submitted 2006-02-06; First posted 2006-02-07 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-05

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm I (Bowman-Birk inhibitor concentrate) (Experimental): Participants are sequentially assigned to 1 of 4 dose level cohorts. One participant in each dose level cohort is randomized to receive placebo. Participants receive 1 of 4 escalating doses of oral Bowman-Birk inhibitor concentrate or placebo, as an orange juice suspension, on day 1.
  Interventions: Drug: Bowman-Birk inhibitor concentrate
- Arm II (placebo) (Placebo Comparator): Participants are sequentially assigned to 1 of 4 dose level cohorts. One participant in each dose level cohort is randomized to receive placebo. Participants receive 1 of 4 escalating doses of oral Bowman-Birk inhibitor concentrate or placebo, as an orange juice suspension, on day 1.
  Interventions: Other: placebo

INTERVENTIONS:
Other: placebo — Given orally
  Other Names: PLCB
  Arms: Arm II (placebo)
Drug: Bowman-Birk inhibitor concentrate — Given orally
  Other Names: BBIC
  Arms: Arm I (Bowman-Birk inhibitor concentrate)

SUMMARY:
This randomized phase I trial is studying the side effects and best dose of Bowman-Birk inhibitor concentrate in preventing cancer in healthy men. Chemoprevention is the use of certain drugs to keep cancer from forming, growing, or coming back. The use of Bowman-Birk inhibitor concentrate may prevent cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the toxic effects of Bowman-Birk inhibitor concentrate, administered as an orange juice suspension, in healthy male participants.

II. Determine a safe dose range of this drug in these participants. III. Determine a recommended phase II dose of this drug in these participants.

SECONDARY OBJECTIVES:

I. Determine the pharmacokinetics of this drug in these participants.

OUTLINE: This is a randomized, placebo-controlled, double-blind, dose-escalation study.

Participants are sequentially assigned to 1 of 4 dose level cohorts. One participant in each dose level cohort is randomized to receive placebo. Participants receive 1 of 4 escalating doses of oral Bowman-Birk inhibitor concentrate or placebo, as an orange juice suspension, on day 1.

After completion of study treatment, participants are followed periodically for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer
* Male
* Performance status - ECOG 0-2
* RBC normal
* WBC ≥ 3,000/mm^3
* Platelet count normal
* Hemoglobin normal
* Hematocrit normal
* ALT and AST normal
* Bilirubin normal
* Creatinine normal
* No history of heart disease
* EKG normal
* No history of pancreatitis or obstruction of pancreatic ducts
* No history of pancreatic cancer or pancreatic adenoma
* Amylase normal
* Lipase normal
* Cholesterol normal
* Triglycerides normal
* Serum glucose ± 10% of normal
* Within 15% of ideal body weight
* No history of chronic medical condition
* No history of excessive alcohol consumption (i.e., > 2 alcoholic beverages per day on average)
* No history of amyloidosis
* Non-smoker

  * Former smokers are eligible provided they have not smoked within the past 3 months
* No history of medical condition that would influence gastrointestinal uptake of the study drug
* No history of diabetes mellitus
* No allergy or prior adverse reaction to soybeans
* Not a vegetarian
* No diagnosis of cancer within the past 5 years except nonmelanoma skin cancer
* No evidence of other life-threatening disease
* No evidence of psychiatric problems
* More than 12 months since prior chemotherapy
* More than 1 month since prior experimental drugs
* More than 3 days since prior consumption of alcoholic beverages
* More than 2 weeks since prior and no concurrent regular use (i.e., > 3 times/week) of nonsteroidal anti-inflammatory drugs
* More than 2 weeks since prior multivitamin tablets (or other vitamin supplements) of > 2 per day
* No more than 2 multivitamin tablets (or other vitamin supplements) per day during study participation
* No more than 1 serving of tofu, soy milk, or other primarily soy-based food per day

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-01; Primary Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Safety as measured by NCI Common Toxicity Criteria and a recommended Phase II dose (RPTD) | Up to 4 weeks

SECONDARY OUTCOMES:
Pharmacokinetics measurements of BBI in the blood and urine | 0 (immediately prior to BBIC administration), 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, and 48 hours after BBIC administration
  Mean, median and 95% confidence interval will then be calculated for each parameter for each dose group. The relationship between dose and the above parameters will be investigated using simple linear regression.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Lustig, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of The University of Pennsylvania, Philadelphia, Pennsylvania, United States